CLINICAL TRIAL: NCT05308797
Title: Comparison of Postoperative Analgesic Efficacy of Combine Serratus Anterior Plane Block and Erector Spinae Plane Block in Coronary Bypass Surgery: Randomized Controlled Study
Brief Title: Combine Serratus Anterior Plane Block Versus Erector Spinae Plane Block in Coronary Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Eda Balcı, Principal investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MH2.4
Record Dates: First submitted 2022-03-18; First posted 2022-04-04 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Cardiac Surgery; Postoperative Pain; Regional Anesthesia Morbidity
Keywords: erector spinae plane block; combined serratus anterior plane block; sternotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): An erector spinae plane block will be performed at the level of the 5th thoracic vertebrae with 30 mL of 0.25% bupivacaine solution under ultrasound guidance before the operation.
  Interventions: Procedure: ESP block
- Combine Serratus Anterior Plane Block (Active Comparator): Combine Serratus Anterior Plane block will be performed at the level of 5th costa with 30 mL of 0.25% bupivacaine (15 mL superficial serratus plane block and 15 mL deep serratus plane block) solution under ultrasound guidance before the operation.
  Interventions: Procedure: CASP block

INTERVENTIONS:
Procedure: ESP block — Preoperative, awake, bilateral, ultrasound-guided erector spinae plane block with 30 mL 0.25 % bupivacaine
  Arms: Erector Spinae Plane Block
Procedure: CASP block — Preoperative, awake, bilateral, ultrasound-guided combine serratus anterior plane block with 30 mL 0.25 % bupivacaine
  Arms: Combine Serratus Anterior Plane Block

SUMMARY:
Even though Erector Spinae Plane (ESP) Block is shown to be efficient in cardiac surgery, the Combine Serratus Anterior Plane (CSAP) Block is still controversial if it has an efficient analgesic effect for sternotomy and drain tube pain relief. This study aims to compare ESP block and CSAP block for postoperative analgesia in coronary bypass surgery patients.

DETAILED DESCRIPTION:
Acute postoperative pain after cardiac surgery originates various surgical procedures that may cause pain including the incision of tissues, sternotomy, the separation of bone-joint structures, the severity and duration of these applications, the use of chest tubes, and the patient's personal inflammatory may affect the response to these stimuli. Postoperative pain is a critical risk factor for the development of pulmonary and cardiovascular complications such as atelectasis, cardiac ischemia, and arrhythmias. Researchers claim that adding techniques to iv drugs, such as thoracic epidural anesthesia, paravertebral block, or erector spinae plane block (ESP) to multimodal analgesia regimens positively affect recovery. Although the efficacy of ESP block in providing postoperative analgesia has been demonstrated in many studies, there is no study comparing CSAP and ESP block in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who will undergo coronary artery bypass grafting surgery with median sternotomy

Exclusion Criteria:

* Emergency surgeries
* Patients with allergic reactions to anesthesia and analgesia drugs to be used
* Patients who do not want to participate in the study voluntarily
* Severe systemic disease (kidney, liver, pulmonary, endocrine)
* Substance abuse history
* History of chronic pain
* Psychiatric problems and communication difficulties
* Patients who need revision due to hemostasis in the postoperative period
* Patients with severe hemodynamic instability due to infection, heavy bleeding, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative 2 hour measurement | 2 hour after ICU admission, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Postoperative 4 hour measurement | 4 hour after ICU admission, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Postoperative 6 hour measurement | 6 hour after ICU admission, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Postoperative 12 hour measurement | 12 hour after ICU admission, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.
Postoperative 24 hour measurement | 24 hour after ICU admission, an average of 5 minutes
  patients will be evaluated in terms of the visual analog pain scale, the scale has a range of 0 to 10. The scale will be shown to patients and 0 means the patient has no pain, 10 means the patient feels the most pain ever felt.

SECONDARY OUTCOMES:
Mechanical ventilation duration | postoperative, approximately 4 to 10 hours
  he total time until patients suitable for endotracheal extubation
Intensive care unit duration | postoperative, approximately 12 to 36 hours
  The total time until patients suitable for discharge from intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: ZELİHA A DEMİR, Professor, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jannati M, Attar A. Analgesia and sedation post-coronary artery bypass graft surgery: a review of the literature. Ther Clin Risk Manag. 2019 Jun 20;15:773-781. doi: 10.2147/TCRM.S195267. eCollection 2019. PMID 31417264
- [Background] Caruso TJ, Lawrence K, Tsui BCH. Regional anesthesia for cardiac surgery. Curr Opin Anaesthesiol. 2019 Oct;32(5):674-682. doi: 10.1097/ACO.0000000000000769. PMID 31356362
- [Background] Jack JM, McLellan E, Versyck B, Englesakis MF, Chin KJ. The role of serratus anterior plane and pectoral nerves blocks in cardiac surgery, thoracic surgery and trauma: a qualitative systematic review. Anaesthesia. 2020 Oct;75(10):1372-1385. doi: 10.1111/anae.15000. Epub 2020 Feb 16. PMID 32062870
- [Background] Abdallah NM, Bakeer AH, Youssef RB, Zaki HV, Abbas DN. Ultrasound-guided continuous serratus anterior plane block: dexmedetomidine as an adjunctive analgesic with levobupivacaine for post-thoracotomy pain. A prospective randomized controlled study. J Pain Res. 2019 Apr 30;12:1425-1431. doi: 10.2147/JPR.S195431. eCollection 2019. PMID 31118760
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Continuous Erector Spinae Plane Block for Rescue Analgesia in Thoracotomy After Epidural Failure: A Case Report. A A Case Rep. 2017 May 15;8(10):254-256. doi: 10.1213/XAA.0000000000000478. PMID 28252539